CLINICAL TRIAL: NCT07330037
Title: A Prospective Phase II Clinical Trial Evaluating Liquid Tumor-infiltrating Lymphocytes (L-TIL) in Combination With Tislelizumab as Adjuvant Therapy in Patients With Resectable Stage II to IIIB (N2) Non-small Cell Lung Cancer (NSCLC) Who Have Undergone Surgery Following Neoadjuvant Treatment With an Immune Checkpoint Inhibitor Plus Platinum-based Doublet Chemotherapy and Did Not Achieve a Pathological Complete Response (pCR)
Brief Title: TALENT Study: Phase II Trial of Adjuvant L-TIL Plus Tislelizumab in Resectable NSCLC Without pCR After Neoadjuvant Chemoimmunotherapy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TALENT
Record Dates: First submitted 2025-12-29; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: NSCLC
MeSH Terms: interventions — tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- L-TIL Cells Plus Tislelizumab (Experimental): Participants will receive adjuvant therapy with liquid tumor-infiltrating lymphocytes (L-TIL) in combination with tislelizumab. Autologous peripheral blood TILs will be infused 4 times, each at a dose of ≥1 × 10⁹ cells, administered 2-3 days after each tislelizumab infusion. Tislelizumab will be given at 400 mg every 6 weeks for a total of 8 cycles of adjuvant treatment.
  Interventions: Biological: L-TIL cells injection; Drug: Tislelizumab

INTERVENTIONS:
Biological: L-TIL cells injection — Autologous peripheral blood TILs will be infused 4 times, each at a dose of ≥1 × 10⁹ cells, administered 2-3 days after each tislelizumab infusion.
Drug: Tislelizumab — Tislelizumab will be given at 400 mg every 6 weeks for a total of 8 cycles of adjuvant treatment.

SUMMARY:
This study evaluates the preliminary efficacy and safety of adjuvant therapy with liquid tumor-infiltrating lymphocytes (L-TIL) in combination with tislelizumab in patients with resectable stage II-IIIB non-small cell lung cancer (NSCLC) who underwent surgery after neoadjuvant treatment with an immune checkpoint inhibitor plus platinum-based doublet chemotherapy but did not achieve a pathological complete response (pCR).

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed NSCLC with imaging indicating resectable stage II-IIIB (N2) disease according to the ninth edition of the AJCC lung cancer TNM staging system;
* No prior anti-tumor treatment;
* Negative for EGFR/ALK/ROS1 mutations;
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0-1;
* Undergone 2-4 cycles of neoadjuvant therapy combining immunotherapy and chemotherapy, followed by surgical resection with R0 margins but without achieving a complete pathological response (non-pCR);
* Adequate organ function as defined below (without using any blood products or hematopoietic growth factors within 14 days):

Normal bone marrow reserve: neutrophil count ≥1.5×10⁹/L, lymphocyte count ≥0.6×10⁹/L, platelet count ≥100×10⁹/L, hemoglobin ≥90g/L; Normal renal function: serum creatinine ≤1.5 mg/dL and/or creatinine clearance rate ≥60 mL/min; Normal liver function: total bilirubin ≤1.5 times ULN, AST and ALT ≤1.5 times ULN; Normal coagulation function: APTT ≤1.5 times ULN, INR ≤1.5 times ULN, PT ≤1.5 times ULN; Left ventricular ejection fraction (LVEF) ≥50% on echocardiography; Pulmonary function test showing FEV1 ≥60%;

* For non-surgically sterilized or women of childbearing potential, must agree to use medically approved contraception (such as an intrauterine device, contraceptive pills, or condoms) during the study treatment period and for 3 months after the end of treatment; must have a negative serum or urine HCG test within 7 days prior to study entry; must not be breastfeeding;

Exclusion Criteria:

* Vaccination within 28 days prior to the first dose, except for inactivated vaccines;
* Major surgery within 28 days prior to the first dose;
* History of other malignancies within 5 years prior to screening;
* Congenital or acquired immunodeficiency, such as HIV infection, or active hepatitis (for inclusion criteria, ALT and AST levels must be within specified limits; for hepatitis B: HBV DNA >10^4/ml; for hepatitis C: HCV RNA >10^3/ml; for chronic hepatitis B carriers, HBV DNA >2000 IU/ml (>10^4 copies/ml), antiviral treatment must be concurrently administered during the study period);
* Unstable or severe concurrent diseases within 6 months prior to the first dose, such as severe/unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction, pulmonary hypertension, life-threatening ventricular arrhythmias requiring maintenance therapy, stroke, and uncontrolled severe seizures;
* Clinically significant active pneumonia or other respiratory system diseases severely affecting lung function at screening;
* Active autoimmune diseases, history of autoimmune diseases, or conditions requiring systemic corticosteroids or immunosuppressive drugs;
* Arterial or venous thrombotic events occurring within 6 months prior to screening;
* History or CT findings indicating active tuberculosis within 1 year prior to enrollment that was untreated;
* Active infections requiring systemic anti-infective treatment;
* Active gastrointestinal bleeding or contraindications to IL-2 use;
* Previous bone marrow transplant or solid organ transplant;
* Other serious acute or chronic medical or psychiatric illnesses (including suicidal ideation or behavior within one year) that may increase the risk associated with participation in the study or administration of the investigational treatment, interfere with the investigational treatment and follow-up, or affect the subject's compliance;

Ages: 17 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
2-year Disease Free Survival | 2 years
  2-year DFS is defined as the proportion of patients who remain free of disease recurrence, second primary malignancy, or death from any cause at 24 months after surgery.

SECONDARY OUTCOMES:
Disease free survival (DFS) | Up to 3 years
  DFS as assessed by the investigator in Stage II- IIIB. DFS defined as the time from the date of randomization to the first observation of disease recurrence (by pathological diagnosis or imaging) or death caused by any reason, whichever occurs first.
Overall survival (OS) | Up to 5 years
  OS defined as the time from the date of randomization to the date of death due to any cause, in Stage II-IIIB and in Stage IB-IIIB
Adverse event (AE) | Up to 5 years
  Incidence and severity of AEs, with severity as determined according to National Cancer Institute Common Terminology Criteria for Adverse Events, version 5.0 (NCI CTCAE v5.0)
Locoregional Recurrence-Free Survival (LRFS) | Up to 3 years
  LRFS was calculated from the date of surgery to the date of first locoregional recurrence; patients without such an event were censored at the date of last follow-up or death.
Distant Metastasis-Free Survival (DMFS) | Up to 3 years
  DMFS was measured from the date of surgery to the date of first distant metastasis; patients without distant metastasis were censored at the last follow-up or at death, whichever occurred first.
Lung Cancer-Specific Survival (LCSS) | Up to 5 years
  Lung cancer-specific survival (LCSS) was calculated from the date of surgery to the date of death due to lung cancer; deaths from other causes were censored at the time of death.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No